CLINICAL TRIAL: NCT01458366
Title: Phase I/II Study of Bendamustine in Combination With Ofatumumab, Carboplatin and Etoposide for Refractory or Relapsed Aggressive B-cell Lymphomas
Brief Title: Phase I/II Study of Bendamustine in Combination With Ofatumumab, Carboplatin and Etoposide
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Collaborators: GlaxoSmithKline (Industry); Novartis (Industry)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 11D.404; 2011-61 (Other: CCRRC); JT 2211 (Other: JeffTrial Number)
Record Dates: First submitted 2011-09-26; First posted 2011-10-24 (Estimated); Results first posted 2020-03-24 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Non-Hodgkin's Lymphoma
Keywords: Non-Hodgkin's Lymphoma; Lymphoma; B-Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma; Lymphoma, B-Cell | interventions — Bendamustine Hydrochloride; ofatumumab; Carboplatin; Etoposide; etoposide phosphate; Tomography Scanners, X-Ray Computed; Magnetic Resonance Spectroscopy; Stem Cell Transplantation; Hematopoietic Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Bendamustine 70mg/m^2 (Experimental): Level 1: Bendamustine 70mg/m^2 Ofatumumab, Carboplatin, and Etoposide
  Interventions: Drug: Bendamustine; Drug: Ofatumumab; Drug: Carboplatin; Drug: Etoposide; Procedure: CT Scan; Procedure: PET Scan; Genetic: Stem Cell Transplant (STC)
- Bendamustine 50mg/m^2 (Experimental): Level -1: Bendamustine 50mg/m^2 Ofatumumab, Carboplatin, and Etoposide
  Interventions: Drug: Bendamustine; Drug: Ofatumumab; Drug: Carboplatin; Drug: Etoposide; Procedure: CT Scan; Procedure: PET Scan; Genetic: Stem Cell Transplant (STC)
- Bendamustine 90mg/m^2 (Experimental): Level 2: Bendamustine 90mg/m^2 Ofatumumab, Carboplatin, and Etoposide
  Interventions: Drug: Bendamustine; Drug: Ofatumumab; Drug: Carboplatin; Drug: Etoposide; Procedure: CT Scan; Procedure: PET Scan; Genetic: Stem Cell Transplant (STC)
- Bendamustine 120mg/m^2 (Experimental): Level 3: Bendamustine 120mg/m^2 Ofatumumab, Carboplatin, and Etoposide
  Interventions: Drug: Bendamustine; Drug: Ofatumumab; Drug: Carboplatin; Drug: Etoposide; Procedure: CT Scan; Procedure: PET Scan; Genetic: Stem Cell Transplant (STC)
- Phase II MTD (Experimental): Phase II: Bendamustine at MTD from Phase I, Ofatumumab, Carboplatin, and Etoposide
  Interventions: Drug: Bendamustine; Drug: Ofatumumab; Drug: Carboplatin; Drug: Etoposide; Procedure: CT Scan; Procedure: PET Scan; Genetic: Stem Cell Transplant (STC)

INTERVENTIONS:
Drug: Bendamustine — Phase 1: Given via IV at the following dose levels:
  * Level 1: 70 mg/m2
  * Level -1: 50 mg/m2
  * Level 2: 90 mg/m2
  * Level 3: 120 mg/m2
  Phase II: Given via IV on Days 1 and 2 of each cycle at the maximum-tolerated dose level found in the Phase I portion of the study.
  Other Names: Ribomustin; Treanda; SDX-105
Drug: Ofatumumab — Phase II
  * Cycle 1: 300 mg via IV on Day 1 and 1000 mg via IV on Day 3
  * Cycles 2 and 3: 1000 mg via IV on Day 1
  Other Names: Arzerra; HuMax-CD20
Drug: Carboplatin — Phase II: AUC 5 via IV on Day 2 of each cycle
  Other Names: cis-Diammine(1,1-cyclobutanedicarboxylato)platinum(II); Paraplatin; Paraplatin-AQ
Drug: Etoposide — Phase II: 100 mg/m2 via IV on Days 1, 2, and 3 of each cycle
  Other Names: Etoposide phosphate; Eposin; Etopophos; Vepesid; VP-16
Procedure: CT Scan — CT Scan to assess disease after Cycle 2 (approximately 25 days) and 3-8 weeks post-treatment
  Other Names: X-ray computed tomography
Procedure: PET Scan — PET Scan to assess disease after Cycle 2 (approximately 25 days) and 3-8 weeks post-treatment
  Other Names: PET; Positron emission tomography
Genetic: Stem Cell Transplant (STC) — For potential transplant candidates:
  * Autologous STC: after 2 cycles of BOCE upon discretion of Thomas Jefferson University hematopoietic stem cell transplant group and in agreement with the study PI or her designee
  * Allogeneic STC: after 2 cycles of BOCE upon discretion of Thomas Jefferson University hematopoietic stem cell transplant group and in agreement with the study PI or her designee
  Other Names: Stem Cell Transplant; Hematopoietic Stem Cell Transplantation; HSCT

SUMMARY:
The Phase I part of the study will apply to identify dose-limiting toxicities (DLT) and to define maximum-tolerated dose (MTD) for a new chemoimmunotherapy combination of bendamustine, ofatumumab, carboplatin, and etoposide in patients with Non Hodgkin's lymphoma whose disease has progressed or has recurred after prior chemotherapy.

The Phase II part of the study will be a single-arm, open-label study in which all patients will receive combination bendamustine, ofatumumab, carboplatin and etoposide at the MTD dose defined in phase I.

This study hopes to identify a life-prolonging therapy for patients with Non-Hodgkin's Lymphoma whose disease has progressed or has recurred after prior chemotherapy. The hypothesis is that the proposed combination of chemotherapy is well-tolerated and is efficacious for the treatment of relapsed/refractory aggressive B cell lymphomas.

DETAILED DESCRIPTION:
Fifty percent of patients with aggressive B cell non-Hodgkin lymphomas are expected to relapse after initial standard chemotherapy. There is no standard salvage regimen for patients with relapsed or refractory disease and at least 75% of patients are expected to succumb to their condition with the commonly used therapy. The recent CORAL study was evaluating the most frequently used rescue regimens R-ICE (rituximab, ifosfamide, carboplatin, etoposide) vs. R-DHAP (rituximab, dexamethasone, high-dose cytarabine and cisplatin) for relapsed aggressive lymphomas, the overall response (OR) was 83% and 3 year event-free survival (EFS) was 47% for "rituximab naïve" patients. In contrast, OR was 51% and 3 year EFS was only 21% in patients who had relapsed after a rituximab containing regimen. There was no significant difference between R-ICE and R-DHAP (in 3-year EFS or overall survival). This study confirmed that rituximab containing rescue was less effective in those patients who had received prior rituximab. Currently, there is virtually no relapsed B-cell lymphoma patients who had not received a rituximab containing induction; therefore, novel strategies are needed to overcome rituximab resistance and to improve overall poor outcome in the relapsed setting. Ofatumumab is a human IgG1 monoclonal anti-CD20 antibody which binds to different CD20 epitopes and is presumed to destroy B cells that are insensitive to rituximab due to their low CD20-expression due to its higher binding avidity and higher antibody and complement dependent cytotoxicity. It was approved by FDA for the treatment of patients with refractory Chronic Lymphocytic Leukemia (CLL). It is being actively studied in low grade and aggressive CD20 positive lymphomas. Bendamustine is an alkylator/purine analogue hybrid cytotoxic compound that has demonstrated single agent activity in lymphomas refractory to other alkylating agents, such as cyclophosphamide. Weidmann et al (2002) demonstrated single agent activity and safety of bendamustine at the dose of 120mg/m2 (day 1, 2) in relapse/refractory aggressive lymphomas. This study had an ORR of 44% in 18 patients. Non-hematological toxicity was mild (13% grade 3 and 0 grade 4). Bendamustine has shown impressive activity and a favorable safety profile when used in combination with rituximab and other cytotoxic drugs: Weide R et al (2007) studied bendamustine (90 mg/m2 day 1, 2) in combination with rituximab and mitoxantrone in 57 patients' with indolent lymphomas and mantle cell lymphoma (MCL). ORR was 92% in follicular and 78% in MCL Vacirca et al presented interim safety analysis of bendamustine (120mg/m2, day 1, 2) and rituximab combination in aggressive B cell lymphomas at 2010 ASCO meeting (in 76 cycles 1 grade 4 neutropenia and 9 additional grade 3 events). Thus, bendamustine combinations are effective and can be given safely in patients with relapsed lymphomas.

The investigators propose a novel R-ICE-like salvage combination regimen in which rituximab is substituted with ofatumumab and ifosfamide with bendamustine in combination with carboplatin and etoposide for refractory or relapsed aggressive B cell lymphomas. The investigators hope to avoid the substantial ifosfamide mediated urinary bladder toxicity (incidence of grade 3 and 4 hemorrhagic cystitis 8-12%) and neurologic toxicity (10-30%: somnolence, confusion, psychosis and seizure) by substituting ifosfamide for bendamustine. The proposed regimen is convenient and can be administered on the outpatient basis which presents an additional benefit to the patients and to the providers. The investigators propose a phase I/II clinical trial and will first determine safety and toxicity of escalating dose bendamustine in combination with fixed doses of ofatumumab, carboplatin and etoposide. The investigators recognize that the commonly used doses of bendamustine in lymphoid malignancies range from 70-120 mg/m2. The investigators will determine maximum-tolerated dose (MTD) and dose-limiting toxicity (DLT) of the combination by using dose escalation of bendamustine from 70mg/m2 in a standard 3 by 3 design. The investigators will then assess efficacy of the combination regimen in relapsed and refractory aggressive B-cell lymphomas.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 and above
2. Patients with histologically confirmed DLBCL, including primary mediastinal large B cell lymphoma, T cell rich B cell lymphoma, "double hit" DLBCL, mantle cell lymphoma, any transformed low grade B cell lymphomas or grade 3 follicular lymphoma (Grade 3a or 3b) who were refractory to RCHOP-like or any anthracycline based chemotherapy or relapsed after at least one prior combination chemotherapeutic regimen and who are deemed candidates for a salvage type chemotherapy.

   * Relapsed disease:
   * Progressive disease after a CR for at least 28 days. Progression will be defined according to the Revised Response Criteria for Malignant Lymphoma (Cheson 2007 (33)).
   * Refractory disease (Subjects must meet one of the following criteria):
   * Persistent or progressive lymphoma with a CR of <28 days duration or with a PR of any duration. Subjects must have received at least 3 cycles of RCHOP-like or any anthracycline base chemotherapy or at least 2 full cycles of HyperCVAD-like chemotherapy.
   * Persistent lymphoma and stable disease after at least 2 cycles of RCHOP-like or any anthracycline base chemotherapy or at least 1 full cycle of HyperCVAD-like chemotherapy (part A and B).
   * Progressive disease despite at least 1 cycle of RCHOP-like or any anthracycline base chemotherapy or at least 1 cycle (part A or A and B) of HyperCVAD-like chemotherapy.
3. Measurable disease, defined by the revised lymphoma criteria (Cheson 2007).
4. Absolute neutrophil count ≥1,500 and platelet count ≥ 75,000, unless due to underlying lymphoma.
5. Left ventricular ejection fraction estimated by MUGA scan or 2D-echocardiogram of at least 45% Cardiology consult is recommended prior to enrollment if a history of coronary artery disease, CHF with estimated LVEF of <50% or clinically significant arrhythmia.
6. Estimated glomerular filtration rate (GFR) must be ≥ 50 mL/min
7. Serum bilirubin ≤ 1.5 × upper limit of normal (ULN) unless deemed elevated secondary to lymphoma involvement of the liver or known Gilbert's syndrome.
8. Aspartate transaminase (AST)/alanine transaminase (ALT) ≤ 2.5 × ULN; unless elevated secondary to lymphoma involvement of the liver
9. Alkaline phosphatase ≤ 2.5 × ULN; unless elevated secondary to lymphoma involvement of the liver.
10. Performance status of ECOG 0-2.
11. Both potentially AutoSCT or AlloSCT candidates and those who are not transplant candidates are eligible for the study.
12. Capable of understanding the investigational nature, potential risks and benefits of the study, and able to provide valid informed consent and HIPAA consent.
13. Female patients of childbearing potential must have a negative serum pregnancy test within 3 days prior to enrollment.
14. Male and female patients of reproductive potential must use an effective contraceptive method during the study and for a minimum of 1 year after the after study treatment.
15. Must be able to comply with study and follow up requirements.

Exclusion Criteria:

1. Current concomitant chemotherapy, radiation therapy, or immunotherapy other than as specified in the protocol.
2. Use of investigational agents within 4 weeks prior to enrollment.
3. Any anticancer therapy within 3 weeks before study entry. The patient must have recovered from all acute toxicities from any previous therapy.
4. Radioimmunotherapy (i.e. Zevalin) within 8 weeks of enrollment.
5. Prior treatment with anti-CD20 monoclonal antibody or alemtuzumab within 4 weeks prior to start of therapy.
6. Autologous stem cell rescue within 12 weeks before study enrollment or those who underwent allogeneic stem cell transplant within one year of enrolment.
7. Known leptomeningeal or parenchymal brain involvement with lymphoma unless in complete remission after treatment for at least 12 weeks with negative CSF cytology within 2 weeks. Prophylaxis of CNS disease using intrathecal dosing of cytotoxic regimens is permitted and should be performed according to the discretion of the treating physician.
8. History of serious organ dysfunction or disease involving the heart, kidney, liver or other organ system that may place the patient at undue risk to undergo treatment.
9. Systemic fungal, bacterial, viral, or other infection if not controlled. Defined as exhibiting ongoing signs/symptoms related to the infection and without improvement, despite appropriate antibiotics or other treatment. (May be enrolled if controlled on treatment).
10. Significant concurrent disease, illness, or psychiatric disorder that would compromise patient safety or compliance, interfere with consent, study participation, follow up, or interpretation of study results.
11. Subjects who have current active hepatic or biliary disease (with exception of patients with Gilbert's syndrome, asymptomatic gallstones, liver metastases or stable chronic liver disease per investigator assessment)
12. History of significant cerebrovascular disease in the past 6 months or ongoing event with active symptoms.
13. Clinically significant cardiac disease including unstable angina, acute myocardial infarction within six months prior to randomization, congestive heart failure (NYHA III-IV), and arrhythmia unless controlled by therapy, with the exception of extrasystoles or minor conduction abnormalities.
14. Other malignancy, unless the patient has been disease-free for at least 3 years following the completion of curative intent therapy, with the following exceptions: treated non-melanoma skin cancer, any in situ carcinoma, or cervical intraepithelial neoplasia, regardless of the disease-free duration, are eligible for this study if definitive treatment for the condition has been completed. Organ-confined prostate cancer with no evidence of recurrent or progressive disease based on prostate-specific antigen (PSA) values are also eligible for this study if hormonal therapy has been initiated, or radical prostatectomy or definitive prostate irradiation has been performed.
15. Positive test for the Human Immunodeficiency Virus (HIV), unless undetectable viral load within 3 months of enrollment (HIV RNA less than 48 copies/mL) on HAART therapy.
16. Positive serology for Hepatitis B (HB) defined as a positive test for HBsAg. . Patients with prior history of Hepatitis B infection, but immune, with only IgG Hepatitis core antibody + (HBcAb +) must be checked for hepatitis B virus titers by PCR and if the viral load is undetectable may be enrolled. These patients must receive anti-viral prophylaxis, such as lamivudine 100 mg po daily (or an equivalent) starting at least one week prior to cycle 1 and continued through the completion of treatment and for 9 months after the last dose of ofatumumab. Hepatitis B virus titers by quantitative PCR and HBsAg should be checked every month (+/- 1 week) while on therapy and every 3 months (+/- 1 month) thereafter for 9 months after the last ofatumumab dose. In the event of an early termination of the clinical trial for any reason, a treating physician will be determining the frequency and the length of follow up studies of hepatitis B virus titers and HBsAg status. It is recommended that the patient remains on prophylactic lamivudine or an equivalent, as above, regardless of whether the study was continued or terminated. In addition, if appropriate consultation with a hepatologist should be obtained.
17. Positive serology for hepatitis C (HC) defined as a positive test for HCAb if confirmed by HC RIBA immunoblot assay (for positive HCAb reflexively perform a HC RIBA immunoblot assay on the same sample)
18. Pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2011-11-09 (Actual); Primary Completion 2018-08-27 (Actual); Study Completion 2020-07-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Filicko-O'Hara, MD, Principal Investigator — Sidney Kimmel Cancer Center at Thomas Jefferson University
Locations (1):
- Sidney Kimmel Cancer Center at Thomas Jefferson University, Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: Kimmel Cancer Center at Thomas Jefferson University, an NCI-Designated Cancer Center — https://www.jeffersonhealth.org/clinical-specialties/cancer
- See also: Thomas Jefferson University Hospitals — http://www.JeffersonHospital.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Bendamustine 70mg/m^2: Combination of Bendamustine, Ofatumumab, Carboplatin, and Etoposide
  Bendamustine:
  - Level 1: 70 mg/m2
- Bendamustine 50mg/m^2: Combination of Bendamustine, Ofatumumab, Carboplatin, and Etoposide
  Bendamustine:
  - Level -1: 50 mg/m2
- Bendamustin 90mg/m^2: Combination of Bendamustine, Ofatumumab, Carboplatin, and Etoposide
  Bendamustine:
  - Level 2: 90 mg/m2
- Bendamustine 120mg/m^2: Combination of Bendamustine, Ofatumumab, Carboplatin, and Etoposide
  Bendamustine:
  - Level 3: 120 mg/m^2
- Bendamustine at MTD: Combination of Bendamustine, Ofatumumab, Carboplatin, and Etoposide
  Bendamustine:
  Phase II at the MTD
Period: Period 1: 70mg/m^2
Arm/Group | Bendamustine 70mg/m^2 | Bendamustine 50mg/m^2 | Bendamustin 90mg/m^2 | Bendamustine 120mg/m^2 | Bendamustine at MTD
Started | 5 | 0 | 0 | 0 | 0
Completed | 3 | 0 | 0 | 0 | 0
Not Completed | 2 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 2 | 0 | 0 | 0 | 0
Period: Period 2: 50mg/m^2
Arm/Group | Bendamustine 70mg/m^2 | Bendamustine 50mg/m^2 | Bendamustin 90mg/m^2 | Bendamustine 120mg/m^2 | Bendamustine at MTD
Started | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Period 3: 90mg/m^2
Arm/Group | Bendamustine 70mg/m^2 | Bendamustine 50mg/m^2 | Bendamustin 90mg/m^2 | Bendamustine 120mg/m^2 | Bendamustine at MTD
Started | 0 | 0 | 3 | 0 | 0
Completed | 0 | 0 | 3 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Period 4: 120mg/m^2
Arm/Group | Bendamustine 70mg/m^2 | Bendamustine 50mg/m^2 | Bendamustin 90mg/m^2 | Bendamustine 120mg/m^2 | Bendamustine at MTD
Started | 0 | 0 | 0 | 3 | 0
Completed | 0 | 0 | 0 | 3 | 0
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Period 5: Maximum Tolerated Dose (MTD)
Arm/Group | Bendamustine 70mg/m^2 | Bendamustine 50mg/m^2 | Bendamustin 90mg/m^2 | Bendamustine 120mg/m^2 | Bendamustine at MTD
Started | 0 | 0 | 0 | 0 | 27
Completed | 0 | 0 | 0 | 0 | 26
Not Completed | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Bendamustine at 50mg/m2 was the dose level -1. No dose limiting toxicities were noted in the first Bendamustine dose level (70mg/m2) so a reduction to 50mg/m2 was not needed and therefore no patients were enrolled at the dose level -1.
Groups:
- Bendamustine 70 mg/m2: Combination of Bendamustine, Ofatumumab, Carboplatin, and Etoposide
  Bendamustine: Phase 1: Given via IV at the following dose levels:
  - Level 1: 70 mg/m2
- Bendamustine 50 mg/m2: Combination of Bendamustine, Ofatumumab, Carboplatin, and Etoposide
  Bendamustine: Phase 1: Given via IV at the following dose levels:
  - Level -1: 50 mg/m2
- Bendamustine 90 mg/m2: Combination of Bendamustine, Ofatumumab, Carboplatin, and Etoposide
  Bendamustine: Phase 1: Given via IV at the following dose levels:
  - Level 2: 90 mg/m2
- Bendamustine 120 mg/m2: Combination of Bendamustine, Ofatumumab, Carboplatin, and Etoposide
  Bendamustine: Phase 1: Given via IV at the following dose levels:
  - Level 3: 120 mg/m2
- Bendamustine at MTD: Combination of Bendamustine, Ofatumumab, Carboplatin, and Etoposide Phase II: Given via IV on Days 1 and 2 of each cycle at the maximum-tolerated dose level found in the Phase I portion of the study.
  Ofatumumab: Phase II
  * Cycle 1: 300 mg via IV on Day 1 and 1000 mg via IV on Day 3
  * Cycles 2 and 3: 1000 mg via IV on Day 1
  Carboplatin: Phase II: AUC 5 via IV on Day 2 of each cycle
  Etoposide: Phase II: 100 mg/m2 via IV on Days 1, 2, and 3 of each cycle
- Total: Total of all reporting groups
Arm/Group | Bendamustine 70 mg/m2 | Bendamustine 50 mg/m2 | Bendamustine 90 mg/m2 | Bendamustine 120 mg/m2 | Bendamustine at MTD | Total
Number analyzed (Participants) | 5 | 0 | 3 | 3 | 27 | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 0 | 3 | 2 | 17 | 24
  >=65 years | 3 | 0 | 0 | 1 | 10 | 14
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1 | 2 | 13 | 17
  Male | 4 | 0 | 2 | 1 | 14 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 5 | 0 | 3 | 3 | 26 | 37
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 1 | 4 | 5
  White | 5 | 0 | 3 | 2 | 20 | 30
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 3 |  | 3 | 3 | 27 | 36

OUTCOME MEASURES:

1. Primary Outcome: Phase I: Maximum-Tolerated Dose of Bendamustine in Combination With Ofatumumab, Carboplatin and Etoposide (BOCE)
Description: To determine the maximum-tolerated dose of bendamustine in combination with ofatumumab, carboplatin and etoposide for patients with refractory or relapsed aggressive B cell lymphomas. Toxicity levels will be assessed after every cycle until a dose-limiting toxicity (DLT) is found. Toxicities will be graded according to the National Cancer Institute Common Terminology Criteria (CTCAE version 4.0). DLT will be defined as any grade 4 infection, or grade >/= 3 non-hematologic toxicity that persists for 7 days or more.
Time Frame: Baseline through 50 days
Population: Patients enrolled on the Phase 1 portion of the study
Measure: Number; unit: mg/m^2
Groups:
- Bendamustine, Ofatumumab, Carboplatin, and Etoposide (BOCE): Combination of Bendamustine, Ofatumumab, Carboplatin, and Etoposide
  Bendamustine: Phase 1: Given via IV at the following dose levels:
  * Level 1: 70 mg/m2
  * Level -1: 50 mg/m2
  * Level 2: 90 mg/m2
  * Level 3: 120 mg/m2
  Phase II: Given via IV on Days 1 and 2 of each cycle at the maximum-tolerated dose level found in the Phase I portion of the study.
  Ofatumumab: Phase II
  * Cycle 1: 300 mg via IV on Day 1 and 1000 mg via IV on Day 3
  * Cycles 2 and 3: 1000 mg via IV on Day 1
  Carboplatin: Phase II: AUC 5 via IV on Day 2 of each cycle
  Etoposide: Phase II: 100 mg/m2 via IV on Days 1, 2, and 3 of each cycle
Arm/Group | Bendamustine, Ofatumumab, Carboplatin, and Etoposide (BOCE)
Number analyzed (Participants) | 11
mg/m^2 | 120

2. Primary Outcome: Overall Frequency of Response With Combination of Bendamustine, Ofatumumab, Carboplatin, and Etoposide at Maximum Tolerated Dose (MTD)
Description: To determine the overall frequency of response with combination bendamustine, ofatumumab, carboplatin, and etoposide for refractory or relapsed aggressive B-cell lymphomas. Overall response is determined as cumulative Complete Response (CR) and Partial Response (PR).
Time Frame: At 25 days and 3-8 weeks post-treatment
Population: Patients who received MTD in phase 1 and the phase 2 patients were evaluated in combined analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Bendamustine, Ofatumumab, Carboplatin, and Etoposide (BOCE)
Number analyzed (Participants) | 28
Participants | 20

3. Secondary Outcome: Phase I: Overall Frequency of Response
Description: To determine the overall frequency of response--overall response will include all subjects with complete response (CR) and partial response (PR). Based on the revised response criteria for malignant lymphoma [Cheson 2007]
  CR= complete disappearance of all detectable clinical evidence of disease and disease related symptoms if present before therapy PR= >/= 50% decrease in sum of the product of the diameters (SPD) of up to 6 of the largest dominant nodes or nodal masses; no increase in size of other nodes, liver or spleen;
Time Frame: CT and PET scans after Cycle 2 (approximately 25 days) and 3-8 weeks post-treatment
Population: For the Phase 1 analysis, participants who received doses of Bendamustine below the MTD were combined for the statistical analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Bendamustine, Ofatumumab, Carboplatin, and Etoposide (BOCE)
Number analyzed (Participants) | 11
Participants | 7

4. Secondary Outcome: Overall Complete Response (CR) and Partial Response (PR) Rate
Description: Based on the revised response criteria for malignant lymphoma [Cheson 2007]
  CR= complete disappearance of all detectable clinical evidence of disease and disease related symptoms if present before therapy PR= >/= 50% decrease in sum of the product of the diameters (SPD) of up to 6 of the largest dominant nodes or nodal masses; no increase in size of other nodes, liver or spleen;
Time Frame: CT and PET scans after Cycle 2 (approximately 25 days) and 3-8 weeks post-treatment
Population: one subject withdrew voluntarily and was not analyzed. The patients enrolled into Phase I portion were combined into one analysis group to compare the two phases of the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Bendamustine, Ofatumumab, Carboplatin, and Etoposide (BOCE)
Number analyzed (Participants) | 35
Participants
  Phase 2: number analyzed (Participants) | 24
  Phase 2: Complete Response | 12
  Phase 2: Partial Response | 4
  Phase 2: No response | 8
  Phase 1: number analyzed (Participants) | 11
  Phase 1: Complete Response | 5
  Phase 1: Partial Response | 3
  Phase 1: No response | 3

5. Secondary Outcome: Overall Progression-Free Survival
Description: To determine 1 and 2 year progression-free survival [Cheson 2007] CR= complete disappearance of all detectable clinical evidence of disease and disease related symptoms if present before therapy PR= >/= 50% decrease in sum of the product of the diameters (SPD) of up to 6 of the largest dominant nodes or nodal masses; no increase in size of other nodes, liver or spleen;
Time Frame: At 1 and 2 years after completion of treatment; year 2 reported
Population: Patients who achieved a complete or partial response. median progression free survival was not achieved in patients undergoing transplant. This population is patients who received the Maximum Tolerated Dose in both Phase I and Phase II. One patient withdrew and was not included in the analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bendamustine, Ofatumumab, Carboplatin, and Etoposide (BOCE)
Number analyzed (Participants) | 28
months | 5.1 [4.0 to NA] — Not enough participants achieved response to calculate upper 95% CI

6. Secondary Outcome: Total Overall Survival for Transplant vs Non-transplant
Description: 1 and 2 year overall survival for those who received Stem Cell Transplant (SCT) versus those who did not receive SCT
Time Frame: At 1 and 2 years after completion of treatment; year 2 reported
Population: One patient withdrew and was not included in the analysis. For the purpose of this analysis, patients in both phases were combined into two groups based on whether or not the patient received a transplant.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bendamustine, Ofatumumab, Carboplatin, and Etoposide (BOCE)
Number analyzed (Participants) | 35
months
  Did not receive transplant | 7.4 [5.7 to NA] — Not enough participants achieved response to calculate upper 95% CI
  Received transplant | 27.3 [26.6 to NA] — Not enough participants achieved response to calculate upper 95% CI

7. Secondary Outcome: Overall Proportion of Patients Who Are Able to Undergo Stem Cell Transplant (SCT)
Description: To determine the proportion of patients who are able to undergo stem cell transplant among transplant-eligible patients. Patients can receive SCT after Cycle 2.
Time Frame: At 2 years after completion of treatment
Population: one subject withdrew voluntarily and was not analyzed. patients from both Phase I and Phase II were analyzed cumulatively for the purpose of analyzing the patients who received a transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Bendamustine, Ofatumumab, Carboplatin, and Etoposide (BOCE)
Number analyzed (Participants) | 35
Participants | 12

8. Secondary Outcome: Overall Safety and Tolerability of the Combination of Bendamustine, Ofatumumab, Carboplatin, and Etoposide
Description: To define safety and tolerability of the combination of ofatumumab, bendamustine, carboplatin and etoposide as measured by the number of dose modifications made to Bendamustine..
  Determined through dose modifications for bendamustine according to patient's toxicity levels:
  * Initial 120 mg/m2 dose decreased to 90 mg/m2
  * Initial 90 mg/m2 dose decreased to 70 mg/m2
  * Initial 70 mg/m2 dose decreased to 50 mg/m2
  * Initial 50 mg/m2 dose decreased to Withdrawn from study
Time Frame: After each cycle (after approximately 3 days, 25 days, and 50 days)
Population: one subject withdrew voluntarily and was not analyzed. As no dose modifications were needed during the study, results of analysis are provided based on the overall patients enrolled to the study.
Measure: Number; unit: dose modifications
Arm/Group | Bendamustine, Ofatumumab, Carboplatin, and Etoposide (BOCE)
Number analyzed (Participants) | 35
dose modifications | 0

ADVERSE EVENTS:
Time Frame: 2 years from baseline
Description: adverse events are presented as a cumulative across both the Phase I and Phase II portions of the study to illustrate the overall safety of the combination of bendamustine, ofatumumab, carboplatin, and etoposide.
Groups:
- Bendamustine at MTD: Phase II: Given via IV on Days 1 and 2 of each cycle at the maximum-tolerated dose level found in the Phase I portion of the study.
  Ofatumumab: Phase II
  * Cycle 1: 300 mg via IV on Day 1 and 1000 mg via IV on Day 3
  * Cycles 2 and 3: 1000 mg via IV on Day 1
  Carboplatin: Phase II: AUC 5 via IV on Day 2 of each cycle
  Etoposide: Phase II: 100 mg/m2 via IV on Days 1, 2, and 3 of each cycle
Arm/Group | Bendamustine 70 mg/m2 | Bendamustine 50 mg/m2 | Bendamustine 90 mg/m2 | Bendamustine 120 mg/m2 | Bendamustine at MTD
All-Cause Mortality (participants affected / at risk) | 4/5 | 0/0 | 1/3 | 1/3 | 16/27
Serious Adverse Events (participants affected / at risk) | 4/5 | 0/0 | 3/3 | 3/3 | 11/27
Other Adverse Events (participants affected / at risk) | 3/5 | 0/0 | 3/3 | 3/3 | 11/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bendamustine 70 mg/m2 (N=5) | Bendamustine 50 mg/m2 (N=0) | Bendamustine 90 mg/m2 (N=3) | Bendamustine 120 mg/m2 (N=3) | Bendamustine at MTD (N=27)
Neutropenic Fever (Blood and lymphatic system disorders) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 4 (5)
thrombocytopenia (Blood and lymphatic system disorders) | 2 (11) | 0 (0) | 2 (13) | 3 (18) | 8 (10)
thromboembolic event (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Hyperglycemia (Blood and lymphatic system disorders) | 1 (8) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hyperkalemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperurecemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (11)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Increase Bilirubin (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 3 (5) | 0 (0) | 2 (5) | 3 (10) | 3 (3)
Decreased ANC (Hepatobiliary disorders) | 3 (5) | 0 (0) | 1 (6) | 3 (7) | 8 (10)
Hypophosphatemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Increased AST (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyponatremia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Decreased ALC (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (17) | 6 (8)
Tumor Lysis Syndrome (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Decreased White Blood Cell Count (Blood and lymphatic system disorders) | 4 (14) | 0 (0) | 3 (7) | 3 (12) | 4 (6)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bendamustine 70 mg/m2 (N=5) | Bendamustine 50 mg/m2 (N=0) | Bendamustine 90 mg/m2 (N=3) | Bendamustine 120 mg/m2 (N=3) | Bendamustine at MTD (N=27)
Anemia (Blood and lymphatic system disorders) | 3 (23) | 0 (0) | 2 (17) | 3 (13) | 11 (17)
Fatigue (General disorders) | 3 (3) | 0 (0) | 2 (2) | 2 (2) | 11 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-17): https://cdn.clinicaltrials.gov/large-docs/66/NCT01458366/Prot_SAP_000.pdf